CLINICAL TRIAL: NCT01984827
Title: A Single Centre, Placebo Controlled, Phase I Study to Evaluate the Effect of Glucose and Moxifloxacin on Cardiac Repolarisation in Male and Female Patients With Type I Diabetes.
Brief Title: Effect of Glucose on QTc Interval in Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Richmond Research Institute (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Organization: Richmond Pharmacology Limited (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RPL-01-12; 2013-001612-30 (EudraCT Number); C12061 (Other: Richmond Pharmacology)
Record Dates: First submitted 2013-11-08; First posted 2013-11-15 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Diabetes
Keywords: Hyperglycaemia; Moxifloxacin; QTc prolongation; C-peptide; Dead in bed syndrome
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia | interventions — Moxifloxacin; Glucose Clamp Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hyper-glycaemic clamp: (Experimental): hyper-glycaemic clamp: intra-venous Glucose as an initial bolus of 250mg/kg followed by a variable maintenance infusion for 4 hours
  Interventions: Other: hyper-glycaemic clamp
- Moxifloxacin (Experimental): Single oral dose of 400 mg Moxifloxacin
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Moxifloxacin — 1. a single oral dose of 400mg Moxifloxacin plus a hyper-glycaemic clamp for 4 hours
  2. a single oral dose of 400mg Moxifloxacin plus C-peptide
  3. a single oral dose of 400mg Moxifloxacin
  4. placebo
  Oral doses of placebo and moxifloxacin will be administered by a Research Physician or Pharmacy staff member between 08:00 a.m. and 10:00 a.m.
  Other Names: Avelox®
  Arms: Moxifloxacin; Placebo
Other: hyper-glycaemic clamp — a hyper-glycaemic clamp only for 2 hours followed by a hyper-glycaemic clamp plus C-peptide for 2 hours
  Other Names: glucose infusion; glucose clamp
  Arms: hyper-glycaemic clamp:

SUMMARY:
High blood glucose levels (hyperglycaemia) and Moxifloxacin (a commonly used antibiotic) have both been shown independently to affect heart activity in healthy volunteers as recorded by ECG. i.e. Both cause prolongation of the QTc interval which is a measure of the time between the start of the Qwave and the end of the Twave during a heartbeat cycle. In this study, the investigators want to find out whether moxifloxacin and hyperglycaemia cause QTc prolongation in Type 1 diabetic patients. The investigators also want to assess whether C-peptide (a fragment if insulin normally found in the blood but not present in the blood of Type 1 diabetics) has the opposite effect on heart activity i.e it shortens the QTc interval will reverse the effect of QTc prolongation in Type 1 diabetes as this may be useful for preventing 'dead in bed' syndrome also known as 'Sudden Cardiac Death' which is more common in diabetic patients compared to healthy volunteers.

DETAILED DESCRIPTION:
The investigators previous research (Taubel et al., 2013) has shown that in healthy individuals glucose by itself can prolong (with C-peptide antagonising the effects) the QT interval, which has long been used as a clinical index of the duration of ventricular repolarisation. This observation warrants serious attention because it suggests that high glucose levels by themselves may be pro-arrhythmogenic. To investigate whether glucose has an effect on cardiac repolarisation, it would be advantageous to test this in an environment uncomplicated by C-peptide. In order to elucidate the effects of glucose on the QTc in the absence of C-peptide, the investigators will use diabetic patients who are no longer able to release endogenous C-peptide. This will allow better understanding to whether (1) the well established QTc prolongation caused by moxifloxacin is exaggerated by elevated levels of blood glucose, which would be important for evaluating the risk in diabetic patients using an IKr blocking drug such as moxifloxacin, and (2) to investigate whether C-peptide substitution will reverse or attenuate the effect in the presence of moxifloxacin. Using the conditions of a formal TQT study, the investigators would also want to confirm the QTc prolonging effects described in Gordin et al. (2008) and whether in this setting C-Peptide substitution will reverse or attenuate the glucose effect on QTc.

This will be a phase I, single centre, randomised, placebo-controlled, open-label, crossover study designed to evaluate the effect of glucose and C-peptide on cardiac repolarisation using a hyperglycaemic clamp and a single 400 mg dose of moxifloxacin as a positive control in non-elderly male and female patients with type I diabetes. The results from this study will form the basis for decisions for future studies.

This study will be performed in compliance with the protocol, ICH GCP and applicable regulatory requirements including EU GMP requirements for investigational medicinal product(s) (IMPs).

ELIGIBILITY:
Inclusion Criteria

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Subject is a male or female with a confirmed diagnosis of C-peptide deficiency Type 1 diabetes mellitus, HbA1c levels of ≤ 60 mmol/mol and 20 - 64 years of age (inclusive) at screening.
2. Healthy (apart from the confirmed diagnosis of C-peptide deficiency Type 1 diabetes mellitus) on the physical examination at screening and at admission on Day -1.
3. Body mass index (BMI) between 18 and 30 kg/m2 (inclusive) at screening and at admission on Day -1, body weight at least 48 kg.
4. Haematology, biochemistry and urinalysis test results within the normal range to a clinically relevant extent at screening and at admission.
5. Female subjects who are either:

   1. Non-childbearing potential, e.g. post-menopausal (as defined as amenorrhoea for at least 12 months with no alternative medical cause) or permanently sterile (permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy) OR
   2. Childbearing potential AND (if heterosexually active) agree to use one or more forms of highly effective contraception as defined below, starting at least one menstrual cycle before first study drug administration and continuing until at least 3 months after the end of the systemic exposure of the study drug.

   Highly effective contraceptive methods for females are as follows:
   * Combined (oestrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation as follows:
   * Oral
   * Intravaginal
   * Transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation as follows:
   * Oral
   * Injectable
   * Implantable
   * Intrauterine device (IUD)
   * Intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion
   * Male partner vasectomised (with documented evidence of azoospermia)
6. Male subjects, if heterosexually active and with a female partner of childbearing potential or a pregnant or breastfeeding partner, must agree to use barrier contraception (male condom) for the treatment period and for at least 3 months after study drug administration. Female partners of male subjects who are of childbearing potential must use one or more forms of highly effective contraception as defined above, starting at least one menstrual cycle before (the male subject's) first study drug administration and continuing until at least 3 months after the last dose of the study drug.

   For male subjects who have had a vasectomy (with documented evidence of azoospermia if possible) and agree to use a barrier method (male condom) for the stated time period, no additional contraceptive method is required by their female partner.
7. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (1996) and applicable regulations, before completing any study-related procedures.
8. Ability to communicate well with the Investigator in the local language, and to understand and comply with the requirements of the study.
9. Subject has a stable diabetic treatment regimen.

Exclusion Criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. History or clinical evidence of Type 1 diabetes mellitus related secondary complications in particular autonomic neuropathy, rhythm disturbances, post medical history of syncope and potassium abnormalities.
2. History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study drug (appendectomy and herniotomy allowed, cholecystectomy not allowed).
3. History or clinical evidence of microvascular disease including chronic kidney failure, macular degeneration or any other disease attributed to the microvascular system that in the Investigator's opinion may affect the outcome of the study.
4. Recent hospitalisation due to hypoglycaemia or hyperglycaemia within the past one month.
5. History of clinically significant syncope.
6. Family history of sudden death.
7. Clinically significant history or family history of congenital long QT syndrome (e.g. Romano-Ward syndrome, Jervell and Lange-Nielson syndrome) or Brugada's syndrome.
8. History of clinically significant arrhythmias and ischemic heart disease (especially ventricular arrhythmias, atrial fibrillation (AF), recent conversion from AF or coronary spasm).
9. Conditions predisposing the volunteer to electrolyte imbalances other than Type 1 diabetes (e.g. altered nutritional states, chronic vomiting, anorexia nervosa, bulimia nervosa).
10. ECG abnormalities in the standard 12-lead ECG (at screening, Day -1 or pre-dose of Day 1) and 24-hour 12 lead Holter ECG or an equivalent assessment and/or submaximal exercise test (at screening) which in the opinion of the Investigator will interfere with the ECG analysis.
11. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes. This includes subjects with any of the following (at screening, Day-1 or pre-dose of Day 1):

    * Sinus node dysfunction.
    * Clinically significant PR (PQ) interval prolongation.
    * Intermittent second or third degree AV block.
    * Incomplete or complete bundle branch block.
    * Sustained cardiac arrhythmia's including (but not limited to) atrial fibrillation or supraventricular tachycardia; any symptomatic arrhythmia with the exception of isolated extra systoles.
    * More than 200 ventricular ectopic beats in 24 hours.
    * Ventricular tachycardia (ventricular tachycardia defined as ≥ 3 successive ventricular ectopic beats at a rate of > 120 bpm).
    * Abnormal T wave morphology.
    * QT interval corrected using the Fridericia's formula (QTcF) > 450 ms. Subject with borderline deviations from these criteria may be included if the deviations do not pose a safety risk, and if agreed between the appointed Cardiologist and the PI.
12. Has vital signs outside of the following normal range at screening, Day -1 or Day 1 predose:

    1. Blood pressure (BP):

       Supine BP (after at least 5 minutes of supine rest):
       * Systolic blood pressure: 90 - 140 mmHg.
       * Diastolic blood pressure: 40 - 90 mmHg.
    2. Supine pulse rate after at least 5 minutes of rest: 45 - 90 bpm.
13. Signs and/or symptoms of a clinically relevant acute illness in the four-week period prior to screening.
14. Veins unsuitable for intravenous puncture or cannulation on either arm (e.g. veins that are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture).
15. Known hypersensitivity to any medicines administered in the trial.
16. Use of prescription medications (other than their usual insulin) within 14 days or 10 half-lives (whichever is longer) prior to Day 1, or any over-the-counter (OTC) medication (including multivitamin, herbal, or homeopathic preparations, excluding hormonal contraception, hormone-replacement therapy, and/or an occasional dose of acetaminophen) within 7 days prior to Day 1 of the dosing period.
17. Administration of antibiotics 7 days prior to the admission for the study or plan to take antibiotics during the study.
18. Treatment with an investigational drug within four weeks prior to admission or having participated in more than three investigational drug studies within one year prior to admission.
19. Positive test results for alcohol or drugs of abuse at screening and on Day -1.
20. Presence or history of drug or alcohol abuse in the last 5 years, or inability to refrain from alcohol use from 48 hours before screening, dosing and each scheduled visit until the end of the study. Alcohol abuse is defined as regular weekly intake of more than 14 units (for both males and females), using the following NHS alcohol tracker http://www.nhs.uk/Tools/Pages/drinks-tracker.aspx.
21. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch, electronic cigarettes) within 3 months prior to the planned first day of dosing.
22. Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening.
23. Has a legal or mental incapacity or language barriers precluding adequate understanding, co-operation, and compliance with the study requirements at screening.
24. Any circumstances or conditions, which, in the opinion of the Investigator, may affect full participation in the study or compliance with the protocol.
25. An inability to follow a standardized diet and meal schedule or inability to fast, as required during the study.
26. Prior screen failure (where the cause of the screen failure is not deemed to be temporary), participation, or enrolment in this study. Subjects who initially failed due to temporary non-medically significant issues are eligible for re-screening once the cause has resolved.
27. Objection by the General Practitioner (GP) to the subject entering the study.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
ECG Analysis | 1, 2, 3 Days
  * The paired PK and QTc interval parameters pre-dose compared to post-administration of glucose. Clinically significant ECG morphology and interval changes from baseline.
  * The effect on QTc will be calculated using concentration-effect analysis.

SECONDARY OUTCOMES:
Proportion of Participants with Adverse Events | 1, 2, 3 Days
  Haematology, chemistry and urinalysis will be used to assess the proportion of subjects with clinically significant changes in laboratory safety tests.
  Electrocardiogram (ECG) will be used to assess the proportion of subjects with morphological heart and/or heart rhythm abnormalities.
  PR, QRS, QT and QTc intervals will be used to assess the proportion of subjects with clinically significant changes in ECG time intervals.
  Systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate and temperature will be used to assess the proportion of subjects with clinically significant changes in vital signs.
  All of the above will be used to measure the incidence of adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, MD FFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd. 1a Newcomen St, London Bridge, London, United Kingdom

REFERENCES:
- [Background] Taubel J, Lorch U, Ferber G, Singh J, Batchvarov VN, Savelieva I, Camm AJ. Insulin at normal physiological levels does not prolong QT(c) interval in thorough QT studies performed in healthy volunteers. Br J Clin Pharmacol. 2013 Feb;75(2):392-403. doi: 10.1111/j.1365-2125.2012.04376.x. PMID 22775199
- [Background] Taubel J, Naseem A, Shakeri-Nejad K, Dingemanse J, Ferber G and Camm A. J. Comparison of digital 12-lead ECG and digital 12-lead holter ECG recordings in healthy male subjects. Clinical Pharmacology and Therapeutics / 89:Supplement 1 (2011) / S11.
- [Derived] Taubel J, Pimenta D, Cole ST, Graff C, Kanters JK, Camm AJ. Effect of hyperglycaemia in combination with moxifloxacin on cardiac repolarization in male and female patients with type I diabetes. Clin Res Cardiol. 2022 Oct;111(10):1147-1160. doi: 10.1007/s00392-022-02037-8. Epub 2022 May 21. PMID 35596784
- See also: Clincal Research Organisation — http://www.richmondpharmacology.com